CLINICAL TRIAL: NCT01183416
Title: High-Dose 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Consolidation of First Remission After Myeloablative Therapy and Autologous Stem-Cell Transplantation in Patients With High-Risk Neuroblastoma: A Phase II Study
Brief Title: High-Dose 3F8/GM-CSF Immunotherapy Plus 13-Cis-Retinoic Acid for Consolidation of First Remission After Myeloablative Therapy and Autologous Stem-Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-158
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2018-10

CONDITIONS: Neuroblastoma
Keywords: GM-CSF; MAB 3F8; RETINOIC ACID (CIS-9 & 13); 09-158
MeSH Terms: conditions — Neuroblastoma | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3F8 monoclonal antibody and 13-cis-Retinoic Acid (Experimental): This phase II, open-label, single arm trial assesses the anti-NB activity of high-dose 3F8 (80 mg/m2/day), which is used in cycles 1-2, with return to standard 3F8 dosage (20 mg/m2/day) in subsequent cycles. The patients are post-transplant and in 1st complete/very good partial remission (CR/VGPR),89 with no evidence of NB by standard studies, but are at high risk for relapse.
  Interventions: Drug: 3F8 monoclonal antibody and 13-cis-Retinoic Acid

INTERVENTIONS:
Drug: 3F8 monoclonal antibody and 13-cis-Retinoic Acid — A cycle consists of treatment with 3F8 for 5 days. GMCSF is started 5 days in advance of each 3F8 cycle. The break between end of a cycle of 3F8/GM-CSF and start of next cycle is 2-to-4-weeks through 4 cycles; subsequent breaks are ~6-8 weeks. 13-cis-retinoic acid is started after cycle 2.

SUMMARY:
The purpose of this study is to see if high-dose 3F8 combined with GM-CSF is better than standard dose 3F8 in treating neuroblastoma. Another purpose of the study is to find out what effects, good and/or bad, 3F8 has on cancer. The investigators also want to see if the antibody works against a very small amount of neuroblastoma (minimal residual disease) that is left in the bone marrow.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NB as defined by a) histopathology (confirmed by the MSKCC Department of Pathology), or b) BM metastases or MIBG-avid lesion(s) plus high urine catecholamine levels.
* High-risk NB as defined by risk-related treatment guidelines1 and the International NB Staging System,89 i.e., stage 4 with (any age) or without (> or = to 18 months of age) MYCN amplification, MYCN-amplified stage 2 or stage 3 (any age), or MYCN-amplified stage 4S.
* The patients are post-stem cell transplantation and in first CR/VGPR, including no measurable MIBG-avid soft tissue tumor assessable for response.
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Creatinine > 3.0 mg/dL
* ALT, AST and Alkaline Phosphatase > 5.0 times the upper limit of normal
* Bilirubin > 3.0 mg/dL
* Patients with grade 3 or higher toxicities (using the CTCAE v3.0) related to cardiac, neurological, pulmonary or gastrointestinal function as determined by physical exam. Patients must have normal blood pressure for age.
* Progressive disease
* History of allergy to mouse proteins.
* Active life-threatening infection.
* Human anti-mouse antibody (HAMA) titer >1000 Elisa units/ml.
* Inability to comply with protocol requirements

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-08; Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kushner BH, Modak S, Basu EM, Roberts SS, Kramer K, Cheung NK. Posterior reversible encephalopathy syndrome in neuroblastoma patients receiving anti-GD2 3F8 monoclonal antibody. Cancer. 2013 Aug 1;119(15):2789-95. doi: 10.1002/cncr.28137. Epub 2013 Apr 30. PMID 23633099
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 4 [3 to 4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Assess the Impact of High-dose 3F8/GM-CSF on Relapse-free Survival
Description: in patients who are post-stem-cell transplantation and in first complete or very good partial remission, but at high risk of relapse.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid
Number analyzed (Participants) | 0

2. Secondary Outcome: Apply Real-time Quantitative RT-PCR to Test the Hypothesis That the Minimal Residual Disease Content of Bone Marrow
Description: after the first treatments with 3F8/GMCSF has significant prognostic impact on relapse-free survival.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid
Number analyzed (Participants) | 0

3. Secondary Outcome: Monitor Safety of the High-dose Antibody Treatment
Description: to assure no side-effects or noxious sequelae develop or emerge that were not seen in the prior phase I study.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid (N=4)
Allergic Reaction (Immune system disorders) | 1
Hypertension (Vascular disorders) | 1
Vacular disorders - Other (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3F8 Monoclonal Antibody and 13-cis-Retinoic Acid (N=4)
Abdominal pain (Gastrointestinal disorders) | 4
Fever (General disorders) | 4
Pain (General disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Urticaria (Skin and subcutaneous tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Edema face (General disorders) | 2
Flushing (Vascular disorders) | 2
Lethargy (Nervous system disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Localized edema (General disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Resp, thoracic & mediastinal disorder Other (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin & subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT01183416/Prot_SAP_000.pdf